CLINICAL TRIAL: NCT04054466
Title: Effectiveness of the Nursing Counseling to the Change of Behavior of Alcohol Consumption in Patients Receiving HAART
Brief Title: Nursing Counseling to the Change of Behavior of Alcohol Consumption in Patients in HAART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); CARIBBEAN, CENTRAL AND SOUTH AMERICA NETWORK FOR HIV EPIDEMIOLOGY (Unknown)
Responsible Party: Principal Investigator, Yesenia Musayon, PhD, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 066991; D43TW009763 (NIH)
Record Dates: First submitted 2019-03-31; First posted 2019-08-13 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: HIV; Alcohol Drinking
Keywords: HIV; Counseling; Antiretroviral Therapy; Alcohol Drinking; Nursing Care
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: The experimentation period will be carried out with a randomized trial type design with concurrent control. The experimental group will receive the counseling and the control group will be constituted by a group of patients randomly selected from the population of patients who started HAART in the last three months in the Strategy who will receive the usual counseling.
  Patients will have a baseline measurement of alcohol consumption, adherence to HAART; then monthly evaluations until six months of intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Intervention with counselling designed
  Interventions: Behavioral: Nursing Counseling in the change of Alcohol Consumption Behavior in patients receiving HAART
- Control group (Other): Intervention with habitual counselling
  Interventions: Behavioral: Habitual Counseling

INTERVENTIONS:
Behavioral: Nursing Counseling in the change of Alcohol Consumption Behavior in patients receiving HAART — It is a health intervention, performed by the nurse with the purpose of providing support or support to the patient's health care. The main objective of counseling is to improve adherence to treatment in patients who receive HAART but also consume alcoholic beverages.
  The components of the differentiated counseling according to the levels of consumption are consolidated according to the recommendations given by the World Health Organization (WHO) after the application of the AUDIT:
  Social consumption (sometime in life, in the last year or in the last month) = mainly education about consumer risks, its application will be bi-monthly.
  Other Names: New Counseling
  Arms: Experimental group
Behavioral: Habitual Counseling — Regular counseling provided to patients receiving HAART, based on education and guidance to comply with antiretroviral treatment
  Other Names: Old Counseling
  Arms: Control group

SUMMARY:
The success of treatment in patients with HIV depends not just on the therapeutic regimen used, but also on the adherence or level of compliance with the treatment achieved by the patient. Patients who consume alcohol are at risk of not complying with antiretroviral treatment, because of the effects caused by alcohol consumption or the interaction that alcohol may have with medications. Differentiated counseling according to consumption levels could help improve the adherence of patients who receive HAART and who also consume alcohol.

The objective of the study is to determine the effectiveness of nursing counseling in improving behavior of alcohol consumption in patients with HIV.

An experimental study will be developed with three phases, and the sampling used in each of the phases will be random.

The first will identify the level of alcohol consumption and adherence to HAART of patients of the Health Strategy of the Hospital Nacional Cayetano Heredia and will develop two focus groups, one with patients and another with nurses to analyze the feasibility, utility, adaptability and Possible effectiveness of the counseling proposed in the improvement of adherence to HAART. In a second phase the intervention will proceed in two groups, one of them is the experimental group where the differentiated counseling will be applied and the second group the control where the habitual counseling will be applied. In the third phase, the counseling undergoing experimentation to evaluate its possible scalability will be subjected again to analysis through focus groups with patients and nurses.

For the evaluation of the variables, different validated instruments will be used: AUDIT for the evaluation of consumption, Simplified Medication Adherence Questionnaire (SMAQ) to assess adherence to HAART, some data will be taken from the patient's clinical history, guides for focus groups will be used.

Descriptive statistics will be used to estimate the level of alcohol consumption and adherence to HAART by patients. The comparability of the study groups in the experimental phase will be evaluated and the effectiveness of the counseling will be demonstrated by comparing means of adherence to HAART before after the intervention.

The project respects the bioethical principles of Charity, Justice and autonomy

DETAILED DESCRIPTION:
Goals:

1. Determine the necessary contents to include the usual counseling to improve the adherence to HAART of patients with HIV according to their different levels of alcohol consumption.
2. To compare the prevalence of alcohol consumption in the last month and last six months between patients who receive and do not receive differentiated nursing counseling according to the level of alcohol consumption.
3. Determine if the intervention is sustainable and scalable.

Material and methods:

Type of study and research design It is an experimental study with three phases, which are detailed below.

First phase The study will start with a formative research to define the content of the intervention strategy, the extension of it, the duration of each session and the approach to be used for each subgroup.

To do this, the level of alcohol consumption of HIV patients receiving HAART and their levels of adherence will first be identified.

Alcohol consumption will be evaluated through the measurement of the prevalence of consumption and the application of the AUDIT (see annex 2) that identifies, alcohol risk consumption, harmful alcohol consumption and dependence. Adherence to HAART will be identified mainly through the SMAQ instrument recommended by the Ministry of Health (see annex 3) for the patients of the strategy and the consistency of this measurement will be sought with the record of the delivery of medications, the treatment card.

Subsequently, the design of the differentiated counseling protocol for the levels of consumption presented by the patients will be concluded. For each component, contents with scientific evidence will be refined. The contrast with the scientific evidence, the available theory and the reality of consumption will consolidate the proposal of counseling.

The elaborated protocol will be submitted to the opinion of focal groups with patients and nurses (see annexes 4 and 5) to validate the proposed counseling and evaluate its usefulness, acceptability, adaptability, feasibility (cost / time), sustainability and possible effectiveness of the proposal. Differentiated counseling for alcohol users according to their consumption levels. Focus groups will be recorded with the prior authorization of the participants.

Finally, the counseling proposal with the feedback received from the focus group will be submitted to the opinion of experts on the subject of HIV, alcohol consumption and nursing counseling. With these tools we will have a counseling protocol (including initial session and follow-up sessions) that will be applied in a pilot test to 10 volunteer patients in order to complete its validation and identify difficulties in its application: 05 patients (for the initial session ) and 05 patients (follow-up session).

Finally, a training program for nurses will be designed in order to have the required profile in the professionals for the application of the counseling.

Second stage Subsequently, the experimentation period will start with a randomized trial type design with concurrent control. The experimental group will receive the counseling and the control group will be constituted by a group of patients randomly selected from the population of patients who started HAART in the last three months in the Strategy who will receive the usual counseling.

Patients will have a baseline measurement of alcohol consumption, adherence to HAART; then monthly evaluations until six months of intervention.

Third phase This final phase will be the analysis of the opinion of patients and nurses on the sustainability (cost / time) scalability of the proposal of differentiated counseling for patients consuming alcohol according to their levels of consumption post experimental evaluation. This phase will be carried out using focus groups: of patients and nurses.

In this phase, the economic evaluation of the intervention will also be carried out. For this purpose, the costs at the market value of all the resources, services or supplies required to carry out the counseling will have been recorded. The cost for each counseling session provided to each patient will also be calculated to then obtain the simple average cost per session for each subgroup according to consumption levels.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to participate in the study.
* Have an assessment of the level of consumption and adherence to HAART.

Exclusion Criteria:

* Have been identified with a level of dependence on alcohol consumption, given that this group of patients requires specialized attention (50).
* Do not consume alcohol.
* Being hospitalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | At the beginning of the study and then every month until the end of six months of follow-up
  Intake of any beverage with alcoholic content reported by the subject throughout his life, last year, last six months, last months and last seven days from an interview, additionally we evaluate Alcohol Disorders through Alcohol Disorders Identification Test (AUDIT).

SECONDARY OUTCOMES:
HAART Adherence | One month after starting antiretroviral treatment and then every month until completing the six months of follow-up.
  Adherence to pharmacological therapy with antiretrovirals is the degree of compliance of the pharmacological treatment according to medical indication and evaluated by the application of the SMAQ. , the record of attendance to the pick up of the medicines and the treatment card.

OTHER OUTCOMES:
Cluster of cuadruple differentiation CD4 T lymphocyte count | Every control made for Hospital until the end of six months of follow-up
  Number of CD4 lymphocytes recorded in the laboratory test performed based on the blood test of the patient receiving HAART, and filed in his Medical Record with the signature of the responsible professional.
Viral load | Every control made for Hospital until the end of six months of follow-up
  Number of replicated copies of the human immunodeficiency virus found per milliliter of blood plasma of the patient receiving HAART and which is recorded in the laboratory result filed in his Medical Record. Said result must be signed by the responsible professional.

CONTACTS AND LOCATIONS:
Overall Officials: Flor Musayón, Dr, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Yesenia Musayón, Lima, Peru

IPD SHARING:
Plan to Share IPD: No
According to the registry of the ethics committee, the study data will only be used for the present investigation.

REFERENCES:
- [Background] Thangavel S, Mulet CT, Atluri VSR, Agudelo M, Rosenberg R, Devieux JG, Nair MPN. Oxidative Stress in HIV Infection and Alcohol Use: Role of Redox Signals in Modulation of Lipid Rafts and ATP-Binding Cassette Transporters. Antioxid Redox Signal. 2018 Feb 1;28(4):324-337. doi: 10.1089/ars.2016.6830. PMID 29132227
- [Background] Dey A, Cederbaum AI. Alcohol and oxidative liver injury. Hepatology. 2006 Feb;43(2 Suppl 1):S63-74. doi: 10.1002/hep.20957. PMID 16447273
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Fishbein M. The role of theory in HIV prevention. AIDS Care. 2000 Jun;12(3):273-8. doi: 10.1080/09540120050042918. PMID 10928203
- [Background] Hankins CA, de Zalduondo BO. Combination prevention: a deeper understanding of effective HIV prevention. AIDS. 2010 Oct;24 Suppl 4:S70-80. doi: 10.1097/01.aids.0000390709.04255.fd. PMID 21042055
- [Background] Baum MK, Rafie C, Lai S, Sales S, Page JB, Campa A. Alcohol use accelerates HIV disease progression. AIDS Res Hum Retroviruses. 2010 May;26(5):511-8. doi: 10.1089/aid.2009.0211. PMID 20455765
- [Background] Room R, Babor T, Rehm J. Alcohol and public health. Lancet. 2005 Feb 5-11;365(9458):519-30. doi: 10.1016/S0140-6736(05)17870-2. PMID 15705462
- [Result] Cook RL, Zhou Z, Kelso-Chichetto NE, Janelle J, Morano JP, Somboonwit C, Carter W, Ibanez GE, Ennis N, Cook CL, Cohen RA, Brumback B, Bryant K. Alcohol consumption patterns and HIV viral suppression among persons receiving HIV care in Florida: an observational study. Addict Sci Clin Pract. 2017 Sep 27;12(1):22. doi: 10.1186/s13722-017-0090-0. PMID 28950912
- [Result] Pokhrel KN, Gaulee Pokhrel K, Neupane SR, Sharma VD. Harmful alcohol drinking among HIV-positive people in Nepal: an overlooked threat to anti-retroviral therapy adherence and health-related quality of life. Glob Health Action. 2018;11(1):1441783. doi: 10.1080/16549716.2018.1441783. PMID 29495948
- [Result] Shuper PA, Neuman M, Kanteres F, Baliunas D, Joharchi N, Rehm J. Causal considerations on alcohol and HIV/AIDS--a systematic review. Alcohol Alcohol. 2010 Mar-Apr;45(2):159-66. doi: 10.1093/alcalc/agp091. Epub 2010 Jan 8. PMID 20061510
- [Result] Chander G, Lau B, Moore RD. Hazardous alcohol use: a risk factor for non-adherence and lack of suppression in HIV infection. J Acquir Immune Defic Syndr. 2006 Dec 1;43(4):411-7. doi: 10.1097/01.qai.0000243121.44659.a4. PMID 17099312
- [Result] Azar MM, Springer SA, Meyer JP, Altice FL. A systematic review of the impact of alcohol use disorders on HIV treatment outcomes, adherence to antiretroviral therapy and health care utilization. Drug Alcohol Depend. 2010 Dec 1;112(3):178-93. doi: 10.1016/j.drugalcdep.2010.06.014. Epub 2010 Aug 11. PMID 20705402
- [Result] Samet JH, Horton NJ, Meli S, Freedberg KA, Palepu A. Alcohol consumption and antiretroviral adherence among HIV-infected persons with alcohol problems. Alcohol Clin Exp Res. 2004 Apr;28(4):572-7. doi: 10.1097/01.alc.0000122103.74491.78. PMID 15100608
- [Result] Cebeci F, Celik SS. Discharge training and counselling increase self-care ability and reduce postdischarge problems in CABG patients. J Clin Nurs. 2008 Feb;17(3):412-20. doi: 10.1111/j.1365-2702.2007.01952.x. Epub 2007 Nov 30. PMID 18047578
- [Result] Kamb ML, Fishbein M, Douglas JM Jr, Rhodes F, Rogers J, Bolan G, Zenilman J, Hoxworth T, Malotte CK, Iatesta M, Kent C, Lentz A, Graziano S, Byers RH, Peterman TA. Efficacy of risk-reduction counseling to prevent human immunodeficiency virus and sexually transmitted diseases: a randomized controlled trial. Project RESPECT Study Group. JAMA. 1998 Oct 7;280(13):1161-7. doi: 10.1001/jama.280.13.1161. PMID 9777816
- [Result] Braithwaite RS, McGinnis KA, Conigliaro J, Maisto SA, Crystal S, Day N, Cook RL, Gordon A, Bridges MW, Seiler JF, Justice AC. A temporal and dose-response association between alcohol consumption and medication adherence among veterans in care. Alcohol Clin Exp Res. 2005 Jul;29(7):1190-7. doi: 10.1097/01.alc.0000171937.87731.28. PMID 16046874
- [Result] Bertholet N, Daeppen JB, Wietlisbach V, Fleming M, Burnand B. Reduction of alcohol consumption by brief alcohol intervention in primary care: systematic review and meta-analysis. Arch Intern Med. 2005 May 9;165(9):986-95. doi: 10.1001/archinte.165.9.986. PMID 15883236
- [Result] Tanner-Smith EE, Lipsey MW. Brief alcohol interventions for adolescents and young adults: a systematic review and meta-analysis. J Subst Abuse Treat. 2015 Apr;51:1-18. doi: 10.1016/j.jsat.2014.09.001. Epub 2014 Sep 16. PMID 25300577
- [Result] Wandera B, Tumwesigye NM, Nankabirwa JI, Mafigiri DK, Parkes-Ratanshi RM, Kapiga S, Hahn J, Sethi AK. Efficacy of a Single, Brief Alcohol Reduction Intervention among Men and Women Living with HIV/AIDS and Using Alcohol in Kampala, Uganda: A Randomized Trial. J Int Assoc Provid AIDS Care. 2017 May/Jun;16(3):276-285. doi: 10.1177/2325957416649669. Epub 2016 May 23. PMID 27215561
- [Result] Noyes ET, Levine JA, Schlauch RC, Crane CA, Connors GJ, Maisto SA, Dearing RL. Impact of Pretreatment Change on Mechanism of Behavior Change Research: An Applied Example Using Alcohol Abstinence Self-Efficacy. J Stud Alcohol Drugs. 2018 Mar;79(2):223-228. doi: 10.15288/jsad.2018.79.223. PMID 29553349
- [Result] Chung MH, Richardson BA, Tapia K, Benki-Nugent S, Kiarie JN, Simoni JM, Overbaugh J, Attwa M, John-Stewart GC. A randomized controlled trial comparing the effects of counseling and alarm device on HAART adherence and virologic outcomes. PLoS Med. 2011 Mar;8(3):e1000422. doi: 10.1371/journal.pmed.1000422. Epub 2011 Mar 1. PMID 21390262
- [Result] Kalichman SC, Grebler T, Amaral CM, McNerey M, White D, Kalichman MO, Cherry C, Eaton L. Intentional non-adherence to medications among HIV positive alcohol drinkers: prospective study of interactive toxicity beliefs. J Gen Intern Med. 2013 Mar;28(3):399-405. doi: 10.1007/s11606-012-2231-1. Epub 2012 Oct 12. PMID 23065532
- See also: Información sobre la medicación y adherencia al tratamiento antirretroviral de gran actividad en pacientes con VIH/SIDA de un hospital de Lima — http://www.scielo.org.pe/scielo.php?script=sci_arttext&pid=S1726-46342015000100010
- See also: Incidence and associated factors to adverse reactions of the initial antiretroviral treatment in patients with HIV — http://www.scielo.org.pe/scielo.php?pid=S1726-46342007000300004&script=sci_abstract&tlng=en
- See also: Análisis de la Situación Epidemiológica del VIH/Sindrome de Inmuno Deficiencia Adquirida (SIDA) en el Perú — http://www.dge.gob.pe/publicaciones/pub_asis/asis19.pdf
- See also: La Dependencia alcohólica como factor de riesgo de tuberculosis multidrogo-resistente — http://cybertesis.unmsm.edu.pe/handle/20.500.12672/2524
- See also: Boletín VIH/Sindrome de Inmuno Deficiencia Adquirida (SIDA) — http://www.dge.gob.pe/portal/docs/vigilancia/vih/Boletin_2015/setiembre.pdf
- See also: Norma Técnica de Salud de Atención Integral del Adulto con Infección por el Virus de la Inmunodeficiencia Humana (VIH) — https://cdn.www.gob.pe/uploads/document/file/187987/187482_R.M_215-2018-MINSA.PDF20180823-24725-6ni25d.PDF
- See also: Principles of Drug Addiction Treatment: A Research-Based Guide — https://www.drugabuse.gov/sites/default/files/podat_1.pdf
- See also: Behavioral counseling after screening for alcohol misuse in primary care: a systematic review and meta-analysis for the US Preventive Services Task Force — https://www.ncbi.nlm.nih.gov/books/NBK109283/
- See also: Treatment for Alcohol Problems: Finding and Getting Help — https://pubs.niaaa.nih.gov/publications/treatment/treatment.htm
- See also: Nutrición y alcoholismo crónico — http://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S0212-16112008000600002